CLINICAL TRIAL: NCT04747873
Title: Investigating the Effectiveness of Incorporating a Stepped Care Approach Into Electronically-delivered CBT for Depression
Brief Title: Incorporating Stepped Care Approach Into e-CBT for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYC-247-21
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Depression; Major Depressive Disorder; Depressive Symptoms
Keywords: Mental Health; Psychotherapy; Depression; Cognitive Behavioural Therapy; Electronic; Internet
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 2 groups. One group will be given 12 weeks of e-CBT for depression. The other group will be given the same 12 weeks of e-CBT modules along with the possibility of additional attention if deemed necessary by the therapist.
Who Masked: Participant
Masking Description: Participants will not be told if they are in a stepped care approach or not. They will all be participating in the same e-CBT modules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-CBT (Experimental): 12 weekly sessions with approximately 30 slides and interactive content, delivered through OPTT designed to mirror in-person standard CBT. Participants go through the content and complete homework at the end of the session. Homework is submitted through OPTT and reviewed by the therapist assigned to the participant, who will provide personalized feedback within three days of submission. Therapists have access to pre-designed session-specific feedback templates to use as a basic structure to write their feedback. By doing so, the time needed to respond to each patient is reduced and therefore the number of patients each therapist can handle increases. On average, developing this feedback takes a therapist 15-20 minutes per patient. In addition to the weekly feedback, participants have the option to message their therapist through the platform throughout the week regarding any questions or concerns they may have.
  Interventions: Behavioral: e-CBT
- e-CBT + Stepped Care (Experimental): 1 - Participant will receive message from assigned care provider on OPTT who check-in with them about strategies and techniques they have discussed and remind them of weekly homework due date.
  2.- Participant will receive phone call from therapist who will check-in on them, remind them of therapy strategies, and verbally remind them of weekly homework due date.
  3 - Participant will receive phone call from assigned care provider who will check-in on them, remind them of some therapy strategies and techniques and weekly session due date, and provide CBT summary of previously reviewed CBT concepts.
  4 - articipant will receive video call (Microsoft Teams) from their therapist who will check-in on them, remind them of weekly session due date, and provide CBT content support to participant.
  5 - Participant will receive CBT sessions in live video call (Microsoft Teams) with research psychiatrist involved in care.
  Interventions: Behavioral: e-CBT; Behavioral: Stepped Care

INTERVENTIONS:
Behavioral: e-CBT — The focus of the sessions is placed on the connection between thoughts, behaviours, emotions, physical reactions, and the environment. We work on evaluating negative beliefs and thought processes and their relationship with depression. Our goal is to adjust the negative thinking so that participants can think about and adapt to the things that are happening to them. This allows them to adjust the way they behave and think about their problems in a way that is not as negative and replaces those thoughts and behaviours with potentially more realistic and productive ones. Participants will be offered e-CBT program over 12 weeks with approximately 30 slides in each module. Participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform.
Behavioral: Stepped Care — Stepped care procedure (see arm/group descriptions).
  Arms: e-CBT + Stepped Care

SUMMARY:
This randomized trial intervention will provide e-CBT for MDD through the Online Psychotherapy Tool (OPTT), a secure, cloud-based, digital mental health platform. Participants (age: 18-65 years) will be offered an e-CBT program tailored to MDD over 12 weeks to address their depressive symptoms. Participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform. The content of the e-CBT modules is designed to mirror in-person standard CBT for MDD. There will be 12 weekly sessions that include approximately 30 slides each along with interactive content, delivered through OPTT. Using clinically validated symptomology questionnaires, the efficacy of the e-CBT program will be evaluated. Both groups will receive the 12-week e-CBT program with one group receiving the standard program. In the second arm, a stepped care approach can be implemented if deemed necessary by the care provider. This decision will be made if the participant has not shown improvement. Questionnaire data along with physiological data will be used to determine the decision.

DETAILED DESCRIPTION:
Participants Participants (n = 110; 55 e-CBT participants, 55 e-CBT + stepped care participants) aged 18-65 years will be recruited at Queen's University from outpatient psychiatry clinic at both Kingston Health Sciences Centre sites (Hotel Dieu Hospital and Kingston General Hospital) as well as Providence Care hospital, family doctors, physicians, clinicians, and self-referrals in Kingston, Ontario, Canada. Once informed consent is provided, participants will be evaluated by a psychiatrist on the research team through secure video appointment to make or confirm a diagnosis of Major Depressive Disorder (MDD) using the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).

The inclusion criteria for the study include the following: at least 18 years of age at the start of the study, diagnosed with major depressive disorder according to DSM-5 by an attending psychiatrist on the research team, competence to consent to participate, ability to speak and read English, and consistent and reliable access to the internet. Exclusion criteria include active psychosis, acute mania, severe alcohol or substance use disorder, and/or active suicidal or homicidal ideation. If a participant is receiving another form of psychotherapy, they will also be excluded from the study, to avoid any confounding effect on the efficacy of this e-CBT program. If eligible for the study, participants will choose between the e-CBT program (n = 55) or the in-person CBT offered individually through this program at Hotel Dieu Hospital (n = 55).

During the informed consent process, it is explained to all participants that this program is not a crisis resource and that they will not have access to their therapist at all times. In the case of an emergency, participants are directed to the proper resources (e.g., emergency department, crisis lines, etc.) and this event will be reported to the principal investigator of the study.

Online Module Content Both e-CBT modules and in-person CBT sessions are designed to instill constructive and balanced coping strategies in participants. During the program, we focus on essential thinking and behavioural skills to help the patients become more engaged in day-to-day activities. The focus of the sessions is placed on the connection between thoughts, behaviours, emotions, physical reactions, and the environment. We work on evaluating negative beliefs and thought processes and their relationship with depression. Our goal is to adjust the negative thinking so that participants can think about and adapt to the things that are happening to them. This allows them to adjust the way they behave and think about their problems in a way that is not as negative and replaces those thoughts and behaviours with potentially more realistic and productive ones.

e-CBT Procedures The e-CBT care plan consists of 12 weekly sessions of approximately 30 slides and interactive content, delivered through OPTT. The e-CBT module content mirrors in-person standard CBT content, including different weekly topics, general information, skill overviews, and homework. Participants are instructed to go through the content and complete homework at the end of the session which helps them practice skills they learned through that session. Homework is submitted through OPTT and reviewed by the therapist assigned to the participant, who will provide personalized feedback within three days of submission. Therapists have access to pre-designed session-specific feedback templates to use as a basic structure to write their feedback. By doing so, the time needed to respond to each patient is reduced and therefore the number of patients each therapist can handle increases. At the same time, by using a structured format in responding to patients, a more standardized quality of care can be assured. The general structure of the feedback template is as follows: -validating the participant's time and effort, -reviewing the event they have used in their homework, -summarizing the previous module's content, and -discussing the participant's homework submission and how they could improve it. In addition to these points, the feedback will have an emphasis on specific content from the participant's submission, reassuring them that their therapist is reading and understanding their challenges. All feedback submissions are finished with a personalized signature from the therapist, helping to develop a rapport between the therapist and the participant. On average, developing this feedback takes a therapist 15-20 minutes per patient. In addition to the weekly feedback, participants have the option to message their therapist through the platform throughout the week regarding any questions or concerns they may have. All technical issues are handled directly through OPTT's technical support team.

Stepped Care Procedure For the stepped care e-CBT group, the decision of whether to add in the additional care will be made starting at the end of week 3. This decision will be made by the principal investigator using the questionnaire and wearable tracker data (Fitbit). The wearable will record heart rate, sleep patterns, and physical activity information. Five possible interventions (see below) may be implemented on a step-by-step basis. If the participant does not show signs of improvement, they will advance to the next step with a total of five steps. Once the participant advances to the next step, they can revert to a previous step if they show signs of improvement or once again advance to the next step if they do not show signs of improvement.

Step 1 (Message from Therapist): The participant will receive a message from their assigned care provider on OPTT who check in with them about some of the strategies and techniques they will have discussed and remind them of their weekly homework due date.

Step 2 (Phone Call): The participant will receive a phone call from their therapist who will check in on them, remind them of some therapy strategies and techniques, and verbally and remind them of their weekly homework due date.

Step 3 (Enhanced Telephone Call): The participant will receive a telephone call from their assigned care provider who will check in on them, remind them of some therapy strategies and techniques and their weekly session due date, and provide a CBT summary of previously reviewed CBT concepts.

Step 4 (Video Call): The participant will receive a video call (via Microsoft Teams) from their therapist who will check in on them, remind them of their weekly session due to date, and provide CBT content support to the participant.

Step 5 (Video Call Sessions): The final stage involves the participant receiving their CBT sessions in a live video call format (via Microsoft Teams) with the research psychiatrist involved in their care.

Training All therapists are research assistants hired by the principal investigator. They all undergo training in psychotherapy and additional training from a psychiatrist on the research team before any interaction with participants. During this training, therapists complete feedback on practice homework, which is reviewed by a psychiatrist on the research team to ensure adequate quality of work. All therapists are supervised by the lead psychiatrist, who is an expert in the area of electronically delivered psychotherapy. Feedback is always reviewed by the lead psychiatrist, before submission to the participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years at the start of the study
* Diagnosis of major depressive disorder according to DSM-5 criteria
* Competence to consent and participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Active psychosis
* Acute mania
* Severe alcohol or substance use disorder
* Active suicidal or homicidal ideation
* Currently receiving another form of psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Change in symptoms (Participant Health Questionnaire - 9 Item) | Week 3, 6, 9, 12
  Clinical standardized symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in symptoms (Quick Inventory of Depressive Symptoms) | Week 1
  Clinical standardized symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire) | Week 1, 6, 12
  Clinical standardized symptom questionnaire. Scale of 1-5, 1 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share results through conference presentations, journal publications, and workshops.
Supporting Information: Study Protocol, SAP
Time Frame: We plan to publish our protocol and statistical analysis plan during the course of the study.
Access Criteria: Participant identification information will always be kept confidential and only anonymized data will be used for the publication of results.

REFERENCES:
- [Derived] Stephenson C, Jagayat J, Kumar A, Khamooshi P, Eadie J, Pannu A, Meartsi D, Danaee E, Gutierrez G, Khan F, Gizzarelli T, Patel C, Moghimi E, Yang M, Shirazi A, Omrani M, Patel A, Alavi N. Comparing clinical decision-making of AI technology to a multi-professional care team in an electronic cognitive behavioural therapy program for depression: protocol. Front Psychiatry. 2023 Dec 21;14:1220607. doi: 10.3389/fpsyt.2023.1220607. eCollection 2023. PMID 38188047
- [Derived] Jagayat JK, Kumar A, Shao Y, Pannu A, Patel C, Shirazi A, Omrani M, Alavi N. Incorporating a Stepped Care Approach Into Internet-Based Cognitive Behavioral Therapy for Depression: Randomized Controlled Trial. JMIR Ment Health. 2024 Feb 9;11:e51704. doi: 10.2196/51704. PMID 38173167
- See also: Publication — https://www-ncbi-nlm-nih-gov.proxy.queensu.ca/pmc/articles/PMC10434487/